CLINICAL TRIAL: NCT04715711
Title: Physiological and Thermoregulatory Responses of Body Cooling During Cycling in a Hot Environment (PYTHON)
Brief Title: Physiological and Thermoregulatory Responses of Body Cooling During Cycling in a Hot Environment
Acronym: PYTHON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: BHSAI (Unknown)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H20-0168
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Participants received four cooling treatments on separate study visits: 1) passive cooling 2) forearm cooling 3) mist-fan cooling, 4) ice towel coolng
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cooling (Active Comparator): Participants will be actively cooled during rest breaks
  Interventions: Other: Forearm coolng; Other: Wet-towel cooling; Other: mist-fan
- No Intervention (Placebo Comparator): Participants will participant in "passive cooling" where they sit in a chair during rest.
  Interventions: Other: passive cooling

INTERVENTIONS:
Other: Forearm coolng — forearm immersion will be performed for active cooling assessment
  Arms: Active Cooling
Other: Wet-towel cooling — Wet towels will be wrapped around the participant's arms for active cooling
  Arms: Active Cooling
Other: mist-fan — a mist-fan will be placed in front of the participant for active cooling
  Arms: Active Cooling
Other: passive cooling — participants will sit in a chair and "passively cool" (no active intervention)
  Arms: No Intervention

SUMMARY:
BHSAI is developing a computational system that provides early alerts of a rise in core body temperature to help reduce the risk of heat injury in the field and during training. The goal of the body temperature alerting system is to use it during rest, exercise in the heat and during body cooling. Using this system during cooling will allow healthcare professionals and military personnel monitor core temperature to ensure cooling is effective (and prevent hypothermia). Therefore, the primary purpose of this investigation is to validate a body temperature alerting system using physiological responses that occur during rest, exercise in the heat and during body cooling. Multiple cooling modalities will be validated. This study is expanding on a previous intervention IRB#H20-0010 (BHSAI Cooling Study), but will examine body cooling during more intense exercise and while cycling. We will also examine the effectiveness of each cooling modality (passive cooling, mist-fan cooling, hand/forearm immersion, ice towel) on physiological variables after exercise in the heat.

DETAILED DESCRIPTION:
Design

The study will be completed in the following timeline:

Visit 1: Baseline and VO2max Testing

Vist 2: Metabolic Heat Production Visit

Visit 3-6: Trial 1, 2 ,3, 4

Visit specific information is described below, however, specific data collection protocols for dependent variables and procedures are included below the description of the study design. Participants will be asked to sign a photo/video release form (Appendix H) to be used in research projects, scientific publications/conferences and for educational purposes. Participants may be videoed or photographed while exercising or resting in the environmental chamber. Participants will be assigned after medical clearance is granted.

Visit 1: Baseline and VO2max Testing

Participants who are approved to participate will be scheduled for a baseline and VO2max testing day. Basal metabolic rate (BMR) will be measured upon arrival during the baseline visit. The participant will lay supine with a ventilated hood covering their head and torso. The ventilated hood will be attached to a hose connected to a metabolic cart. The metabolic cart will continuously measure respiratory exchange ratio, oxygen consumption, and substrate utilization. The participant will remain under the hood for approximately 30 minutes. Upon completion of BMR, participants will provide a urine sample in a clean urine cup. Urine specific gravity and urine color will be assessed. Nude body mass will also be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room. Participants will only be permitted to continue to the VO2max test if the euhydrated criteria of a urine specific gravity (USG) ≤1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status. If USG is greater than 1.025 the subject will be rescheduled for a different day. Height will be measured with a tape measure on Visit 1. Percent body fat will be measured using Air displacement plethysmography (BodPod®; Cosmed, Software Version 4.2+, Concord, CA, USA). This will take less than ~5 minutes to complete. This information will be used to describe the subject demographics. Participants will also be asked to complete a maximal oxygen uptake (VO2max) test on a treadmill and on a cycle ergometer in a thermoneutral environment with about 30 minutes to one hour between. This test will provide aerobic fitness levels of the participants which will be compared between the two exercise protocols. Participants will also be asked about their average weekly physical activity (Appendix K). This visit will take approximately 1-2 hours.

Visit 2: Metabolic Heat Production Visit

In order to prescribe appropriate exercise intensity, heat production must be controlled. Heat production will be prescribed utilizing a graded exercise test (3-5 minute stages) in the heat (same environmental temperature as trials) that will measure metabolic data via collection of expired air utilizing 2-way non-rebreathing mask in order to calculate heat production and appropriately choose cycling intensities to compare between groups of research participants. This test will occur following the baseline visit. The study procedures will mimic those of trials (described below), with the exception of the exercise protocol. The exercise protocol will take approximately 20 minutes to complete. It will include 5 stages of exercise (graded stages). The participant will wear the ACU during this visit.

Visit 3-6: Trials 1-4

Participant numbers will be randomly assigned, and 4 trials (mist-fan, forearm, passive cooling, ice towel) will be ordered with a random number generator and assigned to a participant number.

These orders will be counterbalanced between participants to ensure that there is not an order effect. Each participant will complete four trials as part of the study. Participants will be allowed to make-up trial visits if they are sick, suffer an injury or do not meet hydration requirements. Participants will be asked if they have a current illness or taking medications to determine whether they can complete the exercise trial. The participant's visit will be rescheduled if they have a fever, current illness or taking medications that influence body temperature. Participants will complete four trials on four separate days.

Trial #

Cooling Intervention

1

Passive Cooling

2

Mist-fan Cooling

3

Forearm Immersion

4

Ice Towel

The exercise protocol and recovery portions of this study will be conducted in a climatic chamber with ambient temperature approximately 30-40°C and relative humidity at approximately 30-70%. Participants will drink ad libitum throughout the exercise trial.

Upon arrival to the lab, participants will be asked to indicate if they have consumed alcohol or caffeine in the last 24 hours and 12 hours, respectively. They will not be asked to specify exactly what they have consumed, but if they provide a positive indication, their trial will be rescheduled for another day. Participants will provide a small urine sample in a clean urine cup, and a nude body mass will be measured. Upon arrival to the lab, hydration status will be assessed by urine specific gravity, nude body mass and urine color. Participants will only be permitted to continue to the exercise trial if the euhydrated criteria of a urine specific gravity (USG) ≤1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status. If USG is greater than 1.025 then the subject will be rescheduled for a different day. Participants will be given instructions at the prior visit about how to obtain desired hydration status for the upcoming trial. Researchers will insert an esophageal probe. Only trained personnel are permitted to insert the esophageal probe (no undergraduates will be allowed). Participants will insert a rectal probe and wear a heart rate monitor strap. Additionally, participants will wear 9-site Biopac skin temperature sensors. Researchers will apply the skin temperature sensors with medical tape to the participants' chest, upper arm, forearm, thigh, neck, abdomen, thigh, back, and calf (anterior and posterior). Participants will also wear iButtons (wireless skin temperature sensors) on their chest, upper arm, forearm, thigh, and calf (anterior and posterior). The participants will also be asked to complete a subjective sleep questionnaire upon arriving to the lab. Participants will wear an active combat uniform (ACU) during the exercise trials. Three ADU sizes for the blouse and pants (small, medium, large) will be available for the participants. A belt will be used to ensure the ACU fits appropriately. Participants will not be able to keep the ACU- ADUs will be washed (according to manufacturer's instructions) and re-used for participants. ADU manufacturer's instructions is identical to standard washing cycle (detergent and washing machine dry). The ACU will be weighed before and after use to measure sweat captured in the clothing. Participants will wear the wrist-based devices (provided by BHSAI) on their non-dominant arm throughout the testing. The wrist device must be placed approximately 1-inch proximal to the wrist and be fitted snugly for accurate heart-rate measurements. The wrist device is used to estimate heart rate using infrared technology. The wrist device estimates of heart rate will be compared to the polar heart rate monitor (gold standard). The body alerting system uses heart rate from the wrist device and the environmental conditions to estimate body temperature. The sponsor of the study will use rectal temperature and the 7-site skin temperature sensors to alter the algorithm (not in real time- from the collected data) to better estimate body temperature. The future goal is to have the body alerting system imbedded in the watch. Participants will wear another wrist-based device (WHOOP) on the arm that does not have the BHSAI device. The WHOOP device will monitor heart rate variability and sleep. Participants will be asked to wear this device daily for the duration of the study.

Participants will enter the environmental chamber and sit for 30 minutes to become equilibrated. The environmental chamber will be set to 30-40°C ambient temperature, 30-70% relative humidity After baseline measures of heart rate, rectal temperature, participants will complete the perceptual indices. Participants will also complete an environmental symptoms questionnaire (ESQ).

The trial will consist of two 40-minute intervals of cycling from 7W/kg to 15 W/kg. Each 40-minute exercise block will be followed by a rest break where cooling will occur. Participants will be allowed to drink ad libitum throughout the exercise trial. The participant will be cooled for approximately 30 minutes with their assigned cooling modality. Rectal and esophageal temperature, skin temperature, heart rate, perceptual measures, and mood (POMS, described below) will be collected at various time points before, during, and after exercise and cooling. Metabolic heat production will be measured using indirect calorimetry (mask connected to metabolic cart) during all four trials.

Passive Cooling: Participants will be asked to sit in a chair in the climate chamber for passive cooling.

Mist-fan cooling: A mist-fan will be placed next to the participant and will mist-fan only their hands and forearms during mist-fan cooling. Participants will be asked to roll up their ADU sleeves to increase skin surface area. The temperature of the mist and wind speed of the fan will be recorded.

Forearm immersion: The participant will place their forearm in approximately 20°C water during forearm immersion.

Ice Towel: a towel that can hold water for extended periods will be used and submerged in an ice-water mixture (~2 C). Researchers will gently squeeze the towel to remove excess water (but remain saturated with water) and then apply to both forearms and hands snuggly so that there is no air gap between the towel and the extremity. Apply for 1-5 minutes and then replace it with another fresh, cold towel. This step would ensure that the forearms and hands have near about constant application temperature as the towel would get warm over the application period. The process will be repeated for the entire cooling duration.

Data collection will be divided into two separate phases. A pilot study will be first conducted in which the first two participants will complete all study laboratory visits. Data from those trials will be shared with the sponsor for review before continuation of data collection. Participants will undergo the same procedures for the pilot testing as regular testing. Pilot testing data will be included in the dataset. Following approval from the sponsor, data collection will resume. Each trial will be approximately 4 hours.

All devices will be properly cleaned according to manufacturer's instruction prior to use by other participants.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender man between the ages of 18-28 years
* been cleared by the medical monitor for this study
* VO2max > 45ml/kg/min
* Aerobically active (at least 30 minutes of aerobic exercise 4-5 days per week)

Exclusion Criteria:

* Have a current musculoskeletal injury that would limit their physical activity or preclude the participant from walking, jogging, running, sprinting, or cutting.
* Chronic health problems that affect your ability to thermoregulate (disorders affecting the liver, kidneys or the ability to sweat normally)
* Fever or current illness at the time of testing
* History of cardiovascular, metabolic, or respiratory disease
* A family member died for no apparent reason, had a heart attack, died from heart problems, or sudden death before the age of 50
* Current musculoskeletal injury that limits their physical activity
* Currently taking a medication that is known to influence body temperature (amphetamines, antihypertensives, anticholinergics, acetaminophen, diuretics, NSAIDs, aspirin)
* Identify as cisgender woman, transgender man or transgender woman. Cisgender women, Transgender men, and transgender women are excluded from the current study because the sponsor of the study has requested that this testing be done in physically active cisgender males. It is assumed that they either currently have data on women or transgender women/men to compare this to or have a strategic initiative from a marketing or business perspective that only involves cisgender men.
* Have a history of heat related illness
* Throat or gastroesophageal diseases including gastroesophageal reflux disease (aka, GERD) or difficulty swallowing
* Have any allergies or adverse reactions to the cold (e.g. Cold Uticaria, Raynauds Phenomenon/Disease, or Cryoglobulinanemia)

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Difference in VO2max between Cycle ergometer and treadmill | At the end of exercise test for both cycle ergometer and treadmill
  Participants will be fitted with a Hans Rudolph mask attached to a breathing tube to measure the expired air delivered to the metabolic cart system during the exercise protocol. The metabolic cart will continuously measure oxygen consumption (VO2) to asess their VO2max value.
Metabolic Heat Production | Will be measured continuously throughout the 25 min exercise protocol.
  Participants will be tested for 3-5 minutes at different % of their VO2max. It will include 5 stages.
Change in Rectal Temperature | Measured continuously during two, 40 min exercise blocks and 2 20-30 min cooling periods.
  Rectal thermometer will be self-inserted by participant to assess core temperature
Change in Esophageal Temperature | Measured continuously during two, 40 min exercise blocks and 2 20-30 min cooling periods
  Esophageal thermometer will be inserted by a researcher to assess core temperature
Change in Heart Rate | Measured continuously during two, 40 min exercise blocks and 2 20-30 min cooling periods
  A heart rate monitor will be worn by participant throughout exercise/cooling protocol
Change in Mean Skin temperature | Measured continuously during two, 40 min exercise blocks and 2 20-30 min cooling periods
  Prior to the start of exercise, participants will be instrumented with 9-site (Biopac) and 6-site skin temperature (iButton) sensors. The Biopac skin temperature sensors will be placed on the chest, shoulder, forearm, abdomen, neck, back, thigh and anterior calf and posterior calf. and the iButton skin temperature sensors will be placed on the chest, arm, thigh, and anterior calf and posterior calf.
Change in Rating of Perceived Exertion | Every 10 minutes of the exercise blocks (2 x 40 mins) and cooling period (2 x 20-30 min)
  6-20 scale that indicates how hard the participant feels they are working. 6 represents rest and 20 represents maximal exertion. A high score indicates more perceived exertion.

SECONDARY OUTCOMES:
Change in Thermal Sensation | Every 10 minutes of the exercise blocks (2 x 40 mins) and cooling period (2 x 20-30 min)
  0-8 Scale (cold to hot) that indicated how cold or hot the participate feels. 0 = extremely cold, 8 = extremely hot.
Change in Perception of Fatigue | Every 10 minutes of the exercise blocks (2 x 40 mins) and cooling period (2 x 20-30 min)
  0-10 (no fatigue to extreme fatigue) Scale that indicates how fatigued the participate feels. High score indicates more fatigue (negative outcome).
Change in Perception of thirst | Every 10 minutes of the exercise blocks (2 x 40 mins) and cooling period (2 x 20-30 min)
  0-9 (no thirst to extreme thirst) Scale that indicates how thirsty the subject feels. A higher score is considered a negative outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Korey Stringer Institute, University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No